CLINICAL TRIAL: NCT06156514
Title: Evaluation of Concomitant Chemo-radiotherapy With Cisplatin vs Gemcitabine as the First Line of Treatment in Patients With Locally Advanced Cervical Cancer, With Comorbidities and Preserved Renal Function, is a Phase III Clinical Trial.
Brief Title: Evaluation of Concomitant Chemo-radiotherapy With Cisplatine vs Gemcitabin in Locally Advanced Cervicouterine Cancer
Acronym: MICHELE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, Lucely Cetina Pérez, Principal Investigator, Clinical Professor, National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (018/066/ICI) (CEI/1308/18).
Record Dates: First submitted 2023-06-28; First posted 2023-12-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Cervical Cancer; Gemcitabine; Chemo-radiotherapy
Keywords: Locally advanced cervical cancer (LACC); Concomitant chemo-radiotherapy; Gemcitabine; Cisplatin; Comorbidities
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: This is a phase III clinical trial, open, randomized 1: 1, controlled, noninferiority, in a single hospital center. This study will include 140 patients with the diagnosis of malignant tumors of epithelial origin of the cervix.
  Patients will be randomized 1: 1 to receive in arm "A" (experimental) to receive concomitant chemotherapy based on gemcitabine at 300 mg / m2 weekly and Arm "B" (control) cisplatin 40 mg / m2 weekly, both arms with RT 50.4 Gy in 5 weeks plus 30Gy brachytherapy at the end of the concomitance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Gemcitanine) (Experimental): To receive concomitant chemotherapy based on gemcitabine at 300 mg / m2 weekly
  Interventions: Drug: Gemcitabine
- B (Cisplatin) (Active Comparator): To receive concomitant chemotherapy based on cisplatin 40 mg / m2 weekly
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — Weekly application of gemcitanibe at 300 mg/m2 intravenously in a 30-minute infusion, concomitantly with radiotherapy for a total of 5-6 weeks followed by bachytherapy, in patients diagnosed with locally advanced cervical cancer
  Arms: A (Gemcitanine)
Drug: Cisplatin — Weekly application of Cisplatin at 40 mg/m2 intravenously in a 60-minute infusion, concomitantly with radiotherapy for a total of 5-6 weeks followed by bachytherapy, in patients diagnosed with locally advanced cervical cancer
  Arms: B (Cisplatin)

SUMMARY:
The purpose of this phase III clinical trial, is to evaluate the efficacy and safety of concomitant chemo-radiotherapy with Cisplatin vs Gemcitabine as the first line of treatment in patients with locally advanced cervical cancer, with comorbidities and preserved renal function.

DETAILED DESCRIPTION:
This is a phase III clinical trial, open, randomized 1: 1, controlled, noninferiority, in a single hospital center. This study will include 564 patients with the diagnosis of malignant tumors of epithelial origin of the cervix.

Patients will be randomized 1: 1, arm "A" (experimental) to receive concomitant chemotherapy based on gemcitabine at 300 mg / m2 weekly and Arm "B" (control) to receive cisplatin 40 mg / m2 weekly, both arms with RT 50.4 Gy in 5 weeks plus 30Gy brachytherapy at the end of the concomitance. These patients will be treated in the gynecology-oncology service, candidates for chemo-radiotherapy, it is intended that the recruitment of patients be done in the first 48 months, with a follow-up of 3 years. It is intended to include 3 patients per month, until the total sample is completed in four years. The study is divided into three phases, the first of QT / RT concomitant with gemcitabine or cisplatin depending on the randomized arm; with an approximate duration of 1.5 months with a weekly visit, the second phase is brachytherapy in both arms which lasts from 2 to 7 days, and finally the follow-up phase which lasts for 3 years with a visit every 3 months. In each of the visits we will evaluate the safety of the medication; evaluating adverse events, including laboratory abnormalities as well as acute and chronic toxicity, with the classification according to the common toxicity criteria (CTCAE v4.03) and the efficacy will obtain proportions of clinical and imaging response (TC and / or PET-CT) with the criteria of RECIST v1.1 and / or PERCIST 1.0.

Patient numbers to include. This study will include 140 patients. Test drug, dosage, mode of administration: Gemcitabine at 300 mg / m2 weekly intravenous administration.

Duration of the study 9 years.

ELIGIBILITY:
Inclusion Criteria:

* Singed informed consent.
* Women with Age ≥ 18 years.

  1. -In women of childbearing age it should be documented: a) negative pregnancy test in serum at the beginning of the study (14 days before the start of QT-RT); b) Accept the use of some method of contraception approved by your attending physician during the study and 12 weeks after the treatment has ended.
  2. -In postmenopausal women (surgical or natural menopause) at least one of the following parameters must be met for inclusion.
* Previous bilateral oophorectomy
* Age ≥ 60 years
* Age <60 years and amenorrhea for at least 12 months and levels of follicle stimulating hormone and estradiol within postmenopausal interval parameters.
* Diagnosis of CaCu EC IB2 mg/dl With histological confirmation (epidermoid, adenocarcinoma or adenoescamoso).
* Patients who are candidates for treatment with concomitant QT / RT.
* ECOG 0-2.
* Measurable disease by CT scan and magnetic resonance imaging of the pelvis according to the RECIST criteria v1.1
* No previous treatment.
* Creatinine clearance ≥ 60 ml / min calculated by the CKD-EPI formula.
* Patients with adequate hematological and hepatic functioning, defined by the following parameters:

  1. Hb equal to or greater than 10g /l. (Transfusion prior to treatment is allowed to reach this level of hemoglobin).
  2. Leukocytes greater than or equal to 4000 / mm3.
  3. Platelets equal to or greater than 100,000mm3.
  4. Total bilirubin ≤1.5 times the upper limit of normal (ULN) and. Transaminases less than 1.5 times the LSN
* Patients with a prior diagnosis of the following comorbidities:

  * Diabetes mellitus type 2, which has: fasting serum glucose <250 mg/dl.
  * Systemic arterial hypertension G1 or G2 according to CTCAE v4.03
  * Child Pugh A liver disease
  * Cardiovascular diseases such as: Ischemic heart disease undergoing asymptomatic treatment, without clinical data of stable or unstable angina or for acute myocardial infarction.
  * Compensated heart failure in functional class I of the New York Heart Association.
  * Systemic Lupus Erythematosus with mild or inactive lupus activity (less than or equal to 4 points according to the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI).

Exclusion Criteria:

* Patients with a second neoplasm.
* Pregnant or lactating patients.
* Patients with small cell and / or neuroendocrine CaCu.
* Patients with impaired renal function with a GFR <or equal to 60ml / min calculated by the CKD-EPI formula
* Patients with a history of active TB (TB)
* Patients with a history of Human Immunodeficiency Virus (HIV) infection
* Patients with vesico-vaginal or vesicorectal fistulas at diagnosis
* Concomitant treatment with another experimental drug. Social, family or geographical conditions that suggest a poor attachment to the study

Criteria Interruption of Treatment (Withdrawal of patients)

A patient will be discontinued from the study under the following circumstances:

* Evidence of disease progression.
* If treating physician considers that a change of therapy may benefit the patient.
* If patient withdrew consent
* Due to unmanageable toxicity By pregnancy or if the patient does not wish to continue using the contraceptive methods indicated by the attending physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In the inclusion are patients with the diagnosis confirmed by pathology of cervical-uterine cancer (an exclusive organ of the female gender).
Enrollment: 140 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of concomitant chemoradiotherapy with gemcitabine versus cisplatin in patients with locally advanced cervical cancer (stages IB2-IVA), who have comorbidities and preserved renal function, with progression-free survival rate. | 3 year
  Efficacy will be estimated with progression-free survival: this is defined as the period from the randomization to the first progression documented by imaging studies by RECIST criteria.

SECONDARY OUTCOMES:
To determine the objective response rate after the treatment of concomitant QT-RT with Gemcitabine vs cisplatin in patients with locally advanced cervical cancer with stages IB2-IVA, with comorbidities and preserved renal function. | 8 weeks at the end of treatment
  Objective response rate:
  Percentage of people in a study or treatment group who have a partial or complete response to treatment in a given period of time.
  The measurement is evaluated with RECIST v1.1 or PERCIST criteria
Incidence of Treatment-Emergent Adverse Events of concomitant QT-RT with gemcitabine vs cisplatin in patients with locally advanced cervical cancer with stages IB2-IVA with comorbidities and preserved renal function. | 1 year
  This incidence of Treatment-Emergent Adverse Events will be evaluated through the toxicity profile of the treatment, the evaluation will be classified with the CTCAE v 4.3 criteria.
Determine the Overall Response Rate (ORR) defined as the percentage of people in the study with partial or complete response to treatment in a given period of time, assessed by RECIST v1.1 and PERCIST criteria. | 1 year
  Percentage of people in a study or treatment group who have a partial or complete response to treatment in a given period of time.
  The measurement is evaluated with RECIST v1.1 or PERCIST criteria
  * Complete response as the absence of medible disease.
  * Partial response as the reduction of al least 30% of the size of the tumor (medible disease).
Document the prevalence of comorbidities in this group of patients | Through the study completion, an average of 6 years.
  Point prevalence: refers to the number of cases of a health event at a given time. This is the case to evaluate the presence of comorbidities in patients with cervical cancer at the time of diagnosis of the oncological disease
To evaluate the quality of life of patients with locally advanced cervical cancer with stages IB2-IVA, with comorbidities and preserved renal function with the EORTC QLQ-30. | 1.5 years.
  The quality of life to be evaluated with a given score from 0 to 100, based on the answers of the EORTC QLQ-30 y QLQ Cx-24 questionnaires (patient answer in a 0-4 scale) to the patients at the beginning of treatment, at the fourth week of treatment, during brachytherapy and every three months during the first year of follow up. For symptom scales a high score is indicative of greater problems and for functional scales a low score is indicative of greater problems.
To evaluate the quality of life of patients with locally advanced cervical cancer with stages IB2-IVA, with comorbidities and preserved renal function with the EORTC QLQ CX-24 questionnaires. | 1.5 years.
  The quality of life to be evaluated with a given score from 0 to 100, based on the answers of the EORTC QLQ-30 y QLQ Cx-24 questionnaires (patient answer in a 0-4 scale) to the patients at the beginning of treatment, at the fourth week of treatment, during brachytherapy and every three months during the first year of follow up. For symptom scales a high score is indicative of greater problems and for functional scales a low score is indicative of greater problems.

CONTACTS AND LOCATIONS:
Overall Officials: Eder A Arango, MD, Study Director — National Cancer Institute of Mexico; Lucely C Cetina, MSc, PhD, Principal Investigator — National Cancer Institute of Mexico
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No